CLINICAL TRIAL: NCT01835808
Title: Observational Study of the Evaluation of FFR in the Treatment of Coronary Artery Disease
Brief Title: Portuguese Study on The Evaluation of FFR Guided Treatment of Coronary Disease
Acronym: POST-IT
Status: Completed | Type: Observational
Sponsor: Portuguese Society of Cardiology (Other)
Collaborators: Portuguese Association of Interventional Cardiology (Other); Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: POST-IT
Record Dates: First submitted 2013-04-16; First posted 2013-04-19 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Coronary Artery Disease
Keywords: Fractional flow reserve
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Fractional Flow Reserve: Coronary artery disease patients submitted to coronary angiography and in which coronary lesions are to be evaluated with pressure-wire (FFR functional evaluation).
  Interventions: Device: Fractional flow reserve (St. Jude Medical pressure-wire)

INTERVENTIONS:
Device: Fractional flow reserve (St. Jude Medical pressure-wire) — CAD patients submitted to coronary angiography and in which coronary lesions are to be evaluated with pressure-wire (FFR functional evaluation)
  Other Names: Pressure-Wire (St. Jude Medical)

SUMMARY:
Functional evaluation of coronary lesions, through the evaluation of fractional flow reserve (FFR) with pressure-wire in patients with coronary artery disease (CAD) was evaluated in a randomised trial - the FAME trial - where it was showed to be superior to classic anatomical evaluation. Based on these results, current guidelines recommend the use of FFR (class I-A recommendation) when objective evidence of vessel-related ischemia is not available. Since the FAME trial was published, FFR use increased dramatically in most European countries, Portugal being no exception to this trend. FFR is currently being used in many interventional cardiology centres quite beyond the European Guidelines recommendation, since many physicians now trust more on the information they can collect with pressure-wire during the angiography, and less on non invasive imaging stress tests.

Considering this widespread use of FFR in the evaluation of patients with CAD, there is a need to clarify the clinical results of this approach in a "real patient setting". The Portuguese Study on The Evaluation of FFR Guided Treatment of Coronary Disease (POST-IT) was planned to evaluate if the use of FFR in the decision of coronary revascularization is feasible and allows optimized clinical results in "real world" non selected patients, as showed in clinical randomised trials.

DETAILED DESCRIPTION:
Portuguese Study on The Evaluation of FFR Guided Treatment of Coronary Disease (POST-IT9 is a national multicentric, prospective, consecutive (non selected) anonymous observational study of all patients submitted to coronary angiography and in which functional evaluation with pressure-wire of coronary lesions is to be performed. The main purpose of the registry is to collect data on the medical decisions and clinical results in CAD patients evaluated with FFR (using pressure-wire®, St. Jude Medical), in order to provide evidence in "real world" non selected patients. This evidence will add to the already available clinical data from randomized trials. All Portuguese interventional cardiology centers performing regularly FFR studies were invited to participate in the study. Data will be collected at the time of the procedure and patients will be clinically followed-up for 1 year. Information concerning medical history, past exams, the angiography, the FFR study and the follow-up will be collected on registry forms. The treatment strategy for each patient will be decided by the operator physician, according to his best clinical judgment. Changes in treatment strategy due to FFR results will be recorded, but the intention of the study is just to collect clinical information, and not to influence physician practice. An informed consent form must be signed for all patients included. Patients will be free to withdraw this consent at anytime.

ELIGIBILITY:
Inclusion Criteria:

* consecutive CAD patients submitted to coronary angiography and in which coronary lesions are to be evaluated with pressure-wire (FFR functional evaluation).

Exclusion Criteria:

* Patient not willing to participate (informed consent not signed).
* Life expectancy lower than 12 months (due to cardiac or non-cardiac disease)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive CAD patients submitted to coronary angiography and in which coronary lesions are to be evaluated with pressure-wire (FFR functional evaluation).
Sampling Method: Non-Probability Sample
Enrollment: 918 (Actual)
Dates: Start 2012-03; Primary Completion 2013-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac events | One Year
  Combined endpoint of major adverse cardiac events (cardiovascular mortality, myocardial infarction and coronary revascularization)

SECONDARY OUTCOMES:
Cardiovascular mortality | One Year
  Cardiovascular mortality at one year
Myocardial infarction | One year
  Rate of Myocardial infarction at one year
Coronary revascularization | One year
  Unplanned coronary revascularization at one year

OTHER OUTCOMES:
Impact of FFR in the clinical decision | During the procedure
  Impact (change in the original strategy) of FFR in the clinical decision of interventional cardiologists
Mismatch between non invasive imaging stress tests and FFR | During the procedure
  Mismatch between non invasive imaging stress tests and functional evaluation with FFR in a "real world" (not selected) setting

CONTACTS AND LOCATIONS:
Overall Officials: Sergio B Baptista, MD, Principal Investigator — Hospital Fernando Fonseca, Amadora, Portugal
Locations (1):
- CNCDC, Coimbra, Coimbra District, Portugal

REFERENCES:
- [Derived] Baptista SB, Raposo L, Santos L, Ramos R, Cale R, Jorge E, Machado C, Costa M, Infante de Oliveira E, Costa J, Pipa J, Fonseca N, Guardado J, Silva B, Sousa MJ, Silva JC, Rodrigues A, Seca L, Fernandes R. Impact of Routine Fractional Flow Reserve Evaluation During Coronary Angiography on Management Strategy and Clinical Outcome: One-Year Results of the POST-IT. Circ Cardiovasc Interv. 2016 Jul;9(7):e003288. doi: 10.1161/CIRCINTERVENTIONS.115.003288. PMID 27412867